CLINICAL TRIAL: NCT06917053
Title: Renal Perfusion and the Development of AKI Following Traumatic Injury - A Longitudinal Observational Cohort Study
Brief Title: Renal Perfusion and the Development of AKI Following Traumatic Injury
Acronym: PERTAKI
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 334289
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Haemorrhagic Shock; AKI (Acute Kidney Injury) Due to Trauma; AKI - Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma / serum / urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Traumatic haemorrhagic shock
  Interventions: Device: Ultrasound (including contrast enhanced ultrasound); Device: Sublingual incident dark field videomicroscopy; Device: Urinary oxygen tension.

INTERVENTIONS:
Device: Ultrasound (including contrast enhanced ultrasound) — Ultrasound measures: contrast enhanced ultrasound (CEUS) of the kidney, venous excess ultrasound (VExUS), echocardiography
Device: Sublingual incident dark field videomicroscopy — Sublingual incident dark field (IDF) videomicroscopy
Device: Urinary oxygen tension. — Continuous urinary oxygen tension

SUMMARY:
Acute kidney injury (AKI) is a complication of traumatic haemorrhagic shock (THS) and together these conditions increase mortality risk. Although septic shock patients who develop severe AKI are known to develop hypoperfusion of the renal cortex, little is known regarding intra-renal perfusion changes in THS. The aim of the current study is to investigate the effects of THS on renal microcirculatory perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Within 24 hours of ICU admission following traumatic injury
* Received any blood products during initial resuscitation
* Lactate > 2 mmol/l at any stage prior to study enrolment

Exclusion Criteria:

* Known intolerance to Sonovue or any other ultrasound contrast agent
* Patients with un-survivable injuries / not expected to survive 24 hours in whom the intent of treatment is palliative
* Known CKD 4 or end stage renal failure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to critical care with traumatic haemorrhagic shock who fulfill the inclusion and do no meet any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cortical mean transit time (mTT) measured in seconds | Measured at enrollment, +24 hours and + 48 hours
  Contrast enhanced ultrasound measure of renal cortical tissue blood flow

SECONDARY OUTCOMES:
Cortical perfusion index (PI) measured in arbitrary units | Measured at enrollment, +24 hours and + 48 hours
  Contrast enhanced ultrasound measures of renal cortical tissue blood flow
Cortical wash in rate (WiR) measured in arbitrary units | Measured at enrollment, +24 hours and + 48 hours
  Contrast enhanced ultrasound measures of renal cortical tissue blood flow
Urinary oxygen tension (pO2) across 24 hours study period measured in millimetres of mercury (mmHg) | Across 48 hour study period
  Mean urinary pO2

OTHER OUTCOMES:
Perfused vessel density (PVD) measured in millimetres per square millimetre | Measured at enrollment, +24 hours and + 48 hours
  Incident dark field video microscopy measures of the systemic microcirculation
Microvascular flow index (MFI) (unitless score from 0 to 3 where 3 is the value see in health) | Measured at enrollment, +24 hours and + 48 hours
  Incident dark field video microscopy measures of the systemic microcirculation
Syndecan 1, angiopoietin 1 & 2, Interleukin 6 & 8 (IL-6, IL-8) and tissue necrosis factor (TNF). All measured in nanograms per millilitre (ng/ml) | Measured at enrollment and + 48 hours
  Biomarker analysis - markers of inflammation and endothelial activation/function

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom